CLINICAL TRIAL: NCT07225309
Title: Trial of Meaning Centered Psychotherapy for Mexican Patients With Advanced Cancer
Brief Title: A Study of Meaning-Centered Therapy for Mexican Adults With Advanced Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-240
Record Dates: First submitted 2025-10-15; First posted 2025-11-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer; Thyroid Cancer; Breast Cancer Stage III; Breast Cancer Stage IV; Prostate Cancer Stage III; Prostate Cancer Stage IV; Colorectal Cancer Stage III; Colorectal Cancer Stage IV; Thyroid Cancer Stage III; Thyroid Cancer Stage IV
Keywords: Breast cancer; Breast cancer Stage III; Breast cancer Stage IV; Prostate cancer; Prostate cancer Stage III; Prostate cancer Stage IV; Colorectal cancer; Colorectal cancer Stage III; Colorectal cancer Stage IV; Thyroid cancer; Thyroid cancer Stage III; Thyroid cancer Stage IV; 25-240; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (Experimental): Meaning-Centered Psychotherapy for Latinos (MCP-L)
  Interventions: Behavioral: Meaning-Centered Psychotherapy for Latinos /MCP-L
- Control Intervention (No Intervention): Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Meaning-Centered Psychotherapy for Latinos /MCP-L — MCP-L is a structured 7-session manualized intervention culturally adapted into Spanish for Latino participants diagnosed with advanced cancer, which utilizes a mixture of didactics, discussion and experiential exercises that focus on particular themes related to meaning and advanced cancer. It is 60-minute individual sessions delivered every week or intermittently (depending on participant preference) for up to approximately 3 months (in this time period) in the event of medical illness.
  Arms: Experimental Intervention

SUMMARY:
The purpose of this study is to find out if Meaning-Centered Psychotherapy for Latinos (MCP-L) helps reduce anxiety and depression and improves quality of life compared to cognitive behavioral therapy (CBT). Investigators also want to learn what participants and providers think about the therapy, including how the therapy is designed, outside factors, available resources, and how the people involved affect how well MCP-L works.

ELIGIBILITY:
Patient Eligibility Criteria:

A patient cannot be considered eligible for this study unless ALL of the following conditions are met. Participant eligibility will be determined by an initial EMR review followed by a self-report screener and suicide risk assessment.

Inclusion Criteria:

EMR Criteria

- Documentation of Disease

* Pathologically confirmed breast, prostate, colorectal, or thyroid solid tumor cancer (either most recent or new diagnosis)

  * Definition of Disease [or Measurable Disease]
* Diagnosed with stages III or IV

  * Prior Treatment
* Receiving ambulatory care at INCan

Self-Report Criteria

* Age ≥ 18 years
* Able to read and communicate in Spanish determined by the question: "Can you read and communicate in Spanish? Yes/No"
* Professional role of administrators, clinicians (e.g., oncologists), mental health providers, supervised therapists-in-training (e.g., graduate students), or other related provider delivering the MCP-L experimental intervention
* Providing care (or services) to Mexican cancer patients at INCan
* Has access to internet and an electronic device
* Agrees to be audio-recorded

Exclusion Criteria:

EMR Criteria

* Prior Treatment

  * In the judgment of the treating physician, protocol investigators, and/or study staff, presence of cognitive impairment (e.g., delirium or dementia) sufficient to preclude meaningful informed consent and/or study participation
  * Diagnosed with a major disabling and serious psychiatric condition

Self-Report Criteria

* Presence of suicide risk determined by the Columbia-Suicide Severity Rating Scale
* Too ill to participate determined by the question: "Do you feel too ill to participate because of communication problems, uncontrollable pain, or other symptoms that prevent you from participating?"

Provider Eligibility Criteria:

Inclusion Criteria Self-Report Criteria

* Age ≥ 18 years
* Able to read and communicate in Spanish determined by the question: "Can you read and communicate in Spanish? Yes/No"
* Professional role of administrators, clinicians (e.g., oncologists), mental health providers, supervised therapists-in-training (e.g., graduate students), or other related provider delivering the MCP-L experimental intervention
* Providing care (or services) to Mexican cancer patients at INCan
* Has access to internet and an electronic device
* Agrees to be audio-recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-04-13 (Estimated); Study Completion 2029-04-13 (Estimated)

PRIMARY OUTCOMES:
Change in clinical levels of anxiety and depression for participants participating in Meaning-Centered Psychotherapy for Latinos (MCP-L) | 1 month
  To examine the efficacy of Meaning-Centered Psychotherapy for Latinos (MCP-L) in improving clinical levels of anxiety and depression at 1-month post-intervention follow-up. Assessed using the General Anxiety Disorder 7-item scale (GAD-7; range 0-21, higher scores indicate greater anxiety levels) and the Patient Health Questionnaire 9-item scale (PHQ-9; range 0-27, higher scores indicate greater depression levels), respectively.
Change in clinical levels of anxiety and depression for participants participating in Meaning-Centered Psychotherapy for Latinos (MCP-L) | 3 months
  To examine the efficacy of Meaning-Centered Psychotherapy for Latinos (MCP-L) in improving clinical levels of anxiety and depression at 3-month post-intervention follow-up. Assessed using the General Anxiety Disorder 7-item scale (GAD-7; range 0-21, higher scores indicate greater anxiety levels) and the Patient Health Questionnaire 9-item scale (PHQ-9; range 0-27, higher scores indicate greater depression levels), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Costas Muniz, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Instituto Nacional de Cancerología (INCan), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org